CLINICAL TRIAL: NCT06380374
Title: Evaluation of the Effectiveness of the Program Prepared With Gamification Strategy Based on Multiple Intelligence Theory in Disaster Nursing Education: Randomized Control Study
Brief Title: Gamification in Disaster Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mustafa KILIC, Research Assistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024\01
Record Dates: First submitted 2024-04-02; First posted 2024-04-23 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Gamification; Nursing Students; Multiple Intelligence Theory; Disaster Nursing
Keywords: Gamification; Nursing Students; Multiple Intelligence Theory; Disaster Nursing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamification Group (Experimental): Program Prepared with Gamification Strategy Based on Multiple Intelligence Theory in Disaster Nursing Education
  Interventions: Other: Gamification in Disaster Nursing Education
- Control Group (No Intervention): No intervention was be made to the students in the control group

INTERVENTIONS:
Other: Gamification in Disaster Nursing Education — The contact information of the students who meet the inclusion criteria will be collected by the researchers. The topic of disaster nursing will be explained to all students enrolled in the course by the researcher in the classroom environment. Pre-tests will be taken from students attending the course on disaster nursing. Randomization will be carried out by the researcher, who does not have an active role in the research process. Students in the experimental and control groups will be hidden from the researchers, who will conduct the application until it begins. The Program will be carried out face-to-face. Students in the experimental group will be on the playground. Students will attend the sessions in groups of 6. Each student will compete independently within the group, and each group will have a winner. Students will encounter a total of 30 questions in each game round. The entire game process consists of 7 sessions. After the game process is completed, post-tests will be taken.
  Other Names: Gamification Group
  Arms: Gamification Group

SUMMARY:
This research will be conducted as a randomized controlled study with a parallel design to evaluate the effectiveness of the disaster nursing training program prepared with a gamification strategy based on multiple intelligence theory for final-year public health nursing students. Research hypothesis "H1a: The disaster nursing knowledge level of the students participating in the program, which is prepared with a Gamification Strategy Based on Multiple Intelligence Theory, differs from the control group. H1b: The perception of volunteering towards disaster nursing differs for the students included in the Program Prepared with Gamification Strategy Based on Multiple Intelligence Theory compared to the control group. H1c: The self-efficacy level of students involved in the Program Prepared with Gamification Strategy Based on Multiple Intelligences Theory regarding disaster nursing differs from the control group."

DETAILED DESCRIPTION:
A national study on the subject was used to calculate the research sample size. A study conducted in Turkey determined that students who received training in disaster nursing had a 44% increase in their knowledge level compared to those who did not. In determining the sample size, this ratio is accepted as 95% power and 0.05 alpha level, and the required sample size in the Gpower 3.2 program is 60 people (30 experimental and 30 control). Sampling loss was stated as 17% in another study conducted on a similar population and a similar subject. Students enrolled in the Public Health Nursing course of Selçuk University Faculty of Nursing, the research area, will be evaluated according to the eligibility criteria. Then, the researchers (MK and LS-K) will receive the contact information of the students who meet the inclusion criteria, volunteer to participate in the study, and give consent. The topic of disaster nursing will be explained to all students enrolled in the course by the researcher (LS-K) in the classroom environment. Pre-tests will be taken from students attending the course on disaster nursing by the researchers (MK and LS-K). Randomization will be carried out by the researcher (D-KT), who does not have an active role in the research process. Students in the experimental and control groups will be hidden from the researchers (MK, LS-K, and M-D), who will carry out the application until it begins. The Program prepared for the students in the experimental group, based on the Gamification Strategy Based on Multiple Intelligence Theory, will be carried out face to face. Students in the experimental group will be on the playground. Students will attend the sessions in groups of 6. Each student will compete independently within the group, and each group will have a winner. A total of 30 questions will be encountered in each game round. The entire game process consists of 7 sessions, each expected to last approximately 30 minutes. Post-tests will be taken from the students after the game process is completed. The main result expected from the research is the change in students' knowledge levels about disaster nursing services, their intentions to become volunteer disaster nurses, and their self-efficacy perceptions regarding disaster nursing.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteering to participate in research,
2. Enrollment in the Public Health Nursing course,
3. Not being absent when the subject of disaster nursing is explained.

Exclusion Criteria:

1. Not know to speak Turkish very well,
2. Not volunteering for research,
3. Being an international student,
4. Working as a nurse or healthcare personnel.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Level of knowledge related to disaster nursing services | From enrollment to the end of intervention at 4 weeks
  Knowledge Evaluation Test: Evaluation questions consist of 30 multiple-choice questions and several matching questions. Researchers prepared knowledge assessment questions for disaster nursing education issues. A specification table and scope-matching method were used in its preparation. There is only one correct answer to each question. While creating the Knowledge Assessment Test, expert opinion was taken, and content validity was increased. An increase in the total score indicates that disaster knowledge is high.
Volunteer intention to become a disaster nurse | From enrollment to the end of intervention at 4 weeks
  Two local and three international disaster events were selected to evaluate participants' willingness and perceived ability to respond to different disasters (Covid-19, February 6 Kahramanmaraş earthquake, Töhoku Earthquake and tsunami, Libya Daniel Hurricane and Kastamonu Flood disaster). Students were first asked to mark their willingness to volunteer among options ranging from (1) I am not volunteering, (4) I am volunteering, and then the level of confidence in their abilities, from (1) I am not confident to (4) I am definitely confident in their perceived abilities. The researchers prepared the questions based on the literature
Perception of self-efficacy related to disaster nursing | From enrollment to the end of intervention at 4 weeks
  Disaster Response Self-Efficacy Scale. It consists of a total of 19 items and three sub-dimensions, and the answers were taken on a 5-point Likert scale (1=No self-confidence, 2=basically not self-confident, 3=Somewhat self-confident, 4=Basically self-confident, 5=Full self-confident.). A high score indicates high disaster response self-efficacy. The Cronbach alpha coefficient of the entire scale was determined as 0.96. Cronbach's alpha values for the three dimensions were determined as on-site rescue competence = 0.93, disaster psychological nursing competence = 0.93, and the nature of the role undertaken in the disaster and adaptation competence = 0.93. The three sub-dimensions explain 70.222% of the total variance.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Faculty of Nursing, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: outcomes were used to determine sample size — https://doi.org/10.1016/j.ijdrr.2017.12.008